CLINICAL TRIAL: NCT00708110
Title: A Phase 2a, Multicenter, Randomized, Parallel, Double-Blind, Dose Ranging, Placebo-Controlled Study to Compare Antiviral Effect, Safety, Tolerability and Pharmacokinetics of GSK1349572 Monotherapy Versus Placebo Over 10 Days in HIV-1 Infected Adults (ING111521)
Brief Title: Phase IIa Dose-ranging Study of GSK1349572 in HIV-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111521
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-08

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: dose-ranging study; phase IIa; integrase inhibitor; HIV-1 infection
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Treatment A (Experimental): GSK1349572 2 mg or placebo every 24 hours for 10 days. Screening visit up to 30 days prior to first dose and follow-up for 11 days after last dose.
  Interventions: Drug: GSK1349572; Drug: Placebo
- Treatment B (Experimental): GSK1349572 10 mg or placebo every 24 hours for 10 days. Screening visit up to 30 days prior to first dose and follow-up for 11 days after last dose.
  Interventions: Drug: GSK1349572; Drug: Placebo
- Treatment C (Experimental): GSK1349572 50 mg or placebo every 24 hours for 10 days. Screening visit up to 30 days prior to first dose and follow-up for 11 days after last dose.
  Interventions: Drug: GSK1349572; Drug: Placebo

INTERVENTIONS:
Drug: GSK1349572 — GSK1349572 is an experimental drug being developed for the treatment of HIV. It is in the class of integrase inhibitors.
Drug: Placebo — Placebo is a tablet with no drug in it.

SUMMARY:
GSK1349572 is an integrase inhibitor that will be evaluated for the treatment of HIV infection. This phase IIa, multicenter, randomized, parallel, double-blind, dose ranging, placebo-controlled 'proof of concept' study is to be conducted to compare antiviral effect, safety, tolerability, and pharmacokinetics of GSK1349572 monotherapy versus placebo over 10 days in ART-naïve and experienced, but integrase inhibitor naïve (meaning never having had an integrase inhibitor) HIV-1 infected adults who are not currently receiving antiretroviral therapy. This study consists of a screening visit, a treatment period and a follow-up evaluation. Thirty subjects will be randomized to receive one of three doses of GSK1349572 or placebo q24h over 10 days. Antiviral effect measures include viral load and CD4 cell count.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >/18 and </ 65 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy or bilateral oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study drug.
* CD4+ cell count >/ 100 cells/mm3.
* Documented HIV-1 infection and a screening plasma HIV-1 RNA >/ 5000 copies/mL.
* No current antiretroviral therapy and have not received any in the 12 weeks prior to first dose.
* Capable of giving written informed consent, which includes compliance

Exclusion Criteria:

* The subject has a positive pre-study drug screen. Drugs that will be screened for include amphetamines, barbiturates, cocaine, and PCP.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Prior treatment with an integrase inhibitor (> 1 dose).
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 30 days of study drug administration or anticipated need for such treatment within the study.
* Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (such as hydroxyurea or foscarnet) within 30 days of study drug administration
* Treatment with any vaccine within 30 days prior to receiving study medication.
* Use of multivitamins or antacids within 24 hours prior to the first dose of investigational product.
* History of regular alcohol consumption within 6 months of the screening visit defined as: an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine/serum hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Any condition (including alcohol or drug abuse) which, in the opinion of the investigator, could interfere with the subject's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the subject.
* An active Center for Disease Control and Prevention (CDC) Category C disease [see Appendix 1], except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial.
* History of clinically relevant pancreatitis or hepatitis within the previous 6 months.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
* Has a positive screening Hepatitis B surface antigen; positive screening hepatitis C virus (HCV) antibody and detectable HCV ribonucleic acid (RNA) on subsequent testing. If the hepatitis C antibody is positive but the HCV RNA is undetectable, the subject may be included in the study.
* Inadequate renal function at Screening, defined as either a serum creatinine >1.5 mg/dL or a calculated creatinine clearance (CrCl) ≤ 50 mL/min. A single repeat serum creatinine is allowed to determine eligibility.
* Any acute laboratory abnormality at screen which, in the opinion of the investigator, should preclude the subject's participation in the study of an investigational compound. Any grade 4 laboratory abnormality at screen, with the exception of CPK, will exclude a subject from study participation unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat is allowed for eligibility determination.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3x times the upper limit of normal. A single repeat of ALT and/or AST is allowed for eligibility determination.
* Exclusion Criteria for Screening ECG (A single repeat is allowed for eligibility determination):

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (16):
- United States (16):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Dallas, Texas

REFERENCES:
- [Background] Min S, Sloan L, DeJesus E, Hawkins T, McCurdy L, Song I, Stroder R, Chen S, Underwood M, Fujiwara T, Piscitelli S, Lalezari J. Antiviral activity, safety, and pharmacokinetics/pharmacodynamics of dolutegravir as 10-day monotherapy in HIV-1-infected adults. AIDS. 2011 Sep 10;25(14):1737-45. doi: 10.1097/QAD.0b013e32834a1dd9. PMID 21716073

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received matching placebo tablets orally once daily (QD) for 10 days and were followed for up to 21 days.
- GSK1349572 2 mg QD: Participants received GSK1349572 2 milligram (mg) tablets orally QD for 10 days and were followed for up to 21 days.
- GSK1349572 10 mg QD: Participants received GSK1349572 10 mg tablets orally QD for 10 days and were followed for up to 21 days.
- GSK1349572 50 mg QD: Participants received GSK1349572 50 mg tablets orally QD for 10 days and were followed for up to 21 days.
Period: Overall Study
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Started | 7 | 9 | 9 | 10
Completed | 7 | 9 | 9 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD | Total
Number analyzed (Participants) | 7 | 9 | 9 | 10 | 35
Age Continuous [Mean (Standard Deviation); unit: Years] | 39.6 (10.64) | 41.1 (10.47) | 39.9 (4.14) | 33.7 (10.45) | 38.4 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 9 | 9 | 10 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 2 | 2 | 0 | 3 | 7
  White - White/Caucasian/European Heritage | 5 | 7 | 9 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) at Day 11
Description: Change from Baseline in Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) was calculated as the Day 11 value minus the Baseline value. Blood samples for the measurement of HIV-1 RNA levels were obtained throughout the treatment period (Day 1 to Day 11).
Time Frame: Baseline (Day 1) and Day 11
Population: Intent to Treat Exposed (ITT[E]) Population: all participants who met study criteria and were randomized into the study with documented evidence of having received at least one dose of randomized treatment and at least one post-baseline HIV-1 RNA measurement
Measure: Mean (Standard Deviation); unit: Log10 copies/milliliter (log10 copies/mL
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
Log10 copies/milliliter (log10 copies/mL | 0.05 (0.26) | -1.51 (0.58) | -2.03 (0.49) | -2.46 (0.35)
Statistical Analysis 1: Comparison: Placebo vs GSK1349572 2 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-2.00 to -1.07]
Statistical Analysis 2: Comparison: Placebo vs GSK1349572 10 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-2.52 to -1.55]
Statistical Analysis 3: Comparison: Placebo vs GSK1349572 50 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.48, 95% CI 2-sided [-2.94 to -2.02]

2. Secondary Outcome: Mean Change From Baseline in Plasma HIV-1 RNA to Nadir (Maximum Change) at Day 11
Description: Plasma HIV-1 RNA change from Baseline to the on-treatment nadir (maximum change) was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 11
Population: ITT(E) Population
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
Log10 copies/mL | -0.31 (0.50) | -1.58 (0.55) | -2.09 (0.49) | -2.61 (0.35)

3. Secondary Outcome: Median Change From Baseline in Plasma HIV-1 RNA to Nadir (Maximum Change) at Day 11
Description: as for outcome 2
Time Frame: Baseline and Day 11
Population: ITT(E) Population
Measure: Median (Full Range); unit: Log10 copies/mL
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
Log10 copies/mL | -0.12 [-1.39 to 0.00] | -1.65 [-2.34 to -0.86] | -1.99 [-2.71 to -1.43] | -2.55 [-3.28 to -2.16]

4. Secondary Outcome: Plasma HIV-1 RNA Rate of Decline Over 10 Days
Description: The rate of decline of plasma HIV-1 RNA levels from Day 1 to Day 11 was measured.
Time Frame: Day 1 to Day 11
Population: ITT(E) Population
Measure: Mean (90% Confidence Interval); unit: Log10 copies/mL/day
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
Log10 copies/mL/day | 0 [-0.01 to 0.01] | -0.14 [-0.16 to -0.12] | -0.20 [-0.21 to -0.18] | -0.25 [-0.27 to -0.24]

5. Secondary Outcome: Number of Participants With HIV-1 RNA <400 Copies/mL and <50 Copies/mL
Description: The number of participants who achieved plasma HIV-1 RNA levels <400 copies/mL and <50 copies/mL through Day 11 was measured.
Time Frame: Day 11
Population: ITT(E) Population
Measure: Number; unit: participants
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
participants
  <400 copies/mL | 0 | 1 | 4 | 9
  <50 copies/mL | 0 | 1 | 0 | 4

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) and Over 24 Hours (AUC[0-24]) of GSK1349572 Following Dose Administration on Day 1
Description: AUC is defined as the area under the GSK1349572 concentration-time curve as a measure of drug exposure. AUC(0-inf) is defined as the area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time. AUC(0-24) is defined as the area under the concentration-time curve from time zero (pre-dose) to24 hours. Blood samples for pharmacokinetic (PK) analysis of GSK1349572 were obtained on Day 1at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration.
Time Frame: Day 1
Population: Pharmacokinetic Summary (PKS) Population: participants (par.) with an evaluable profile of GSK1349572 on Day 10. Par. were excluded if they vomited within 2 hours of dosing on Day 10, missed more than one dose 2 days prior to Day 10, and took prohibited concomitant medication during the treatment period. No par. were analyzed in the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms*hour per milliliter (µg*hr/mL
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
Micrograms*hour per milliliter (µg*hr/mL
  AUC(0-inf) |  | 2.63 (39) | 10.1 (26) | 40.5 (33)
  AUC(0-24) |  | 2.05 (33) | 7.41 (27) | 30.34 (33)

7. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) and Concentration at 24 Hours Post Dose (C24) of GSK1349572 Following Dose Administration on Day 1
Description: Cmax is defined as the maximum observed plasma concentration, and C24 is defined as the concentration at 24 hours post dose. Blood samples for PK analysis of GSK1349572 were obtained on Day 1at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration. From the plasma concentration-time curve, Cmax was determined by standard non-compartmental analysis using WinNonlin Pro 4.1 or higher.
Time Frame: Day 1
Population: PKS Population. No participants were analyzed in the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (µg/mL)
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
Micrograms per milliliter (µg/mL)
  Cmax |  | 0.18 (35) | 0.57 (28) | 2.46 (32)
  C24 |  | 0.03 (49) | 0.15 (30) | 0.59 (31)

8. Primary Outcome: Time to Maximum Observed Concentration (Tmax) and Absorption Lag Time (Tlag) of GSK1349572 Following Dose Administration on Day 1
Description: tmax is defined as the time to the maximum obsevered plasma concentration. Absorption lag time is defined as the time taken for a drug to appear in the systemic circulation following administration. tlag was estimated based on PK sampling times of 0 (pre-dose), 0.5, 1, 1.5, 2 3, 4, 6, 8, 12, and 24 hours post-dose. Blood samples for PK analysis of GSK1349572 were obtained on Day 1at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration. From the plasma concentration-time curve, tmax was determined by standard non-compartmental analysis using WinNonlin Pro 4.1 or higher.
Time Frame: Day 1
Population: PKS Population. No participants were analyzed for the placebo group.
Measure: Median (Full Range); unit: Hours
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
Hours
  tmax |  | 1.50 [0.50 to 3.00] | 2.00 [1.02 to 6.00] | 2.09 [1.00 to 3.97]
  tlag |  | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

9. Primary Outcome: Terminal Half-life (t1/2) of GSK1349572 Following Dose Administration on Day 1
Description: The terminal half-life (t1/2) of GSK1349572 is defined as the time required for the plasma concentration of GSK1349572 to reach half of its original concentration. Blood samples for PK analysis of GSK1349572 were obtained on Day 1at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration.
Time Frame: Day 1
Population: PKS Population. No participants were analyzed for the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
Hours |  | 10.7 (30) | 11.8 (22) | 11.2 (29)

10. Primary Outcome: Apparent Clearance (CL/F) of GSK1349572 Following Dose Administration on Day 1
Description: The CL/F is defined as the apparent total clearance of the drug from plasma after oral administration. Blood samples for PK analysis of GSK1349572 were obtained on Day 1at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration.
Time Frame: Day 1
Population: PKS Population. No participants were analyzed for the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/hr)
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
Liters per hour (L/hr) |  | 0.76 (39) | 0.99 (26) | 1.23 (33)

11. Primary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC[0-tau]) of GSK1349572 Following the Last Repeat Administration on Day 10
Description: AUC is defined as the area under the GSK1349572 concentration-time curve as a measure of drug exposure. AUC(0-tau) is defined as the area under the concentration-time curve over the dosing interval. Blood samples for PK analysis of GSK1349572 were obtained on Day 10at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration.
Time Frame: Day 10
Population: PKS Population. No participants were analyzed for the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
µg*hr/mL |  | 2.56 (29) | 10.13 (20) | 43.39 (20)

12. Primary Outcome: Pre-dose Concentration (C0), Concentration at the End of the Dosing Interval (Ctau), Minimum Observed Concentration During One Dosing Interval (Cmin), and Maximum Obsevered Plasma Concentration (Cmax) of GSK1349572 Following the Last Repeat Administration
Description: C0 is defined as the pre-dose concentration. Ctau is defined as the concentration at the end of the dosing interval. Cmin is defined as the minimum observed concentration during one dosing interval. Cmax is defined as the maximum obsevered plasma concentration. Blood samples for PK analysis of GSK1349572 were obtained on Day 10 at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration.
Time Frame: Day 10
Population: PKS Population. No participants were analyzed for the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
µg/mL
  C0 |  | 0.04 (51) | 0.20 (28) | 0.82 (44)
  Ctau |  | 0.04 (50) | 0.19 (25) | 0.83 (26)
  Cmin |  | 0.04 (51) | 0.19 (26) | 0.81 (43)
  Cmax |  | 0.22 (25) | 0.80 (23) | 3.34 (16)

13. Primary Outcome: Time to the Maximum Observed Concentration (Tmax) of GSK1349572 Following the Last Repeat Administration on Day 10
Description: tmax is defined as the time to the maximum obsevered plasma concentration. Blood samples for PK analysis of GSK1349572 were obtained on Day 10 at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration. From the plasma concentration-time curve, tmax was determined by standard non-compartmental analysis using WinNonlin Pro 4.1 or higher.
Time Frame: Day 10
Population: PKS Population. No participants were analyzed for the placebo group.
Measure: Median (Full Range); unit: Hours
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
Hours |  | 1.00 [0.42 to 3.00] | 1.48 [0.50 to 3.00] | 2.00 [0.97 to 4.00]

14. Primary Outcome: Terminal Half-life (t1/2) of GSK1349572 Following the Last Repeat Administration on Day 10
Description: The terminal half-life (t1/2) of GSK1349572 is defined as the time required for the plasma concentration of GSK1349572 to reach half of its original concentration. Blood samples for PK analysis of GSK1349572 were obtained on Day 10 at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration.
Time Frame: Day 10
Population: PKS Population. No participants were analysed for the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
Hours |  | 11.13 (24) | 11.64 (21) | 11.95 (22)

15. Primary Outcome: Apparent Clearance (CL/F) of GSK1349572 Following Dose Administration on Day 10
Description: The CL/F is defined as the apparent total clearance of the drug from plasma after oral administration. Blood samples for PK analysis of GSK1349572 were obtained on Day 10 at pre-dose (within 15 minutes prior to dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post GSK1349572 dose administration.
Time Frame: Day 10
Population: PKS Population. No participants were analyzed for the placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 0 | 9 | 7 | 10
L/hr |  | 0.78 (29) | 0.99 (20) | 1.15 (20)

16. Primary Outcome: Number of Participants With Any Non-serious Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From Baseline (Day 1) until Follow-up (average of 3 study weeks)
Population: Safety Population: all participants who were randomized into the study with documented evidence of having received at least one dose of randomized treatment
Measure: Number; unit: participants
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
participants
  Any Non-serious AE | 5 | 4 | 7 | 7
  Any SAE | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants Who Received the Indicated Concomitant Medications During the Study Period
Description: Concomitant medications received during the study period are presented by generic term. Only those concomitant medications that were received by at least two participants are presented. "Multiple ingredient" is the term used in the statistical package for items that contain more than one active ingredient.
Time Frame: From Baseline (Day 1) until Follow-up (average of 3 study weeks)
Population: Safety Population. Only those participants who received a concomitant medication were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 5 | 4 | 9 | 10
participants
  Multiple ingredients (combination product) | 3 | 2 | 4 | 5
  Ibuprofen | 0 | 0 | 3 | 2
  Bupropion hydrochloride | 0 | 1 | 1 | 1
  Escitalopram oxalate | 2 | 0 | 1 | 0
  Acetylsalicylic acid | 0 | 1 | 0 | 1
  Ascorbic acid | 1 | 1 | 0 | 0
  Cyanocobalamin | 0 | 1 | 1 | 0
  Fish oil | 0 | 0 | 1 | 1
  Loratadine | 0 | 0 | 2 | 0
  Ranitidine hydrochloride | 0 | 0 | 1 | 1
  Trazodone | 0 | 0 | 1 | 1
  Valacyclovir hydrochloride | 1 | 0 | 0 | 1
  Vitamin B substances (not otherwise specified) | 1 | 0 | 0 | 1
  Zolpidem tartrate | 0 | 0 | 1 | 1

18. Primary Outcome: Change From Baseline in Mean Blood Pressure at Days 1, 4, 7, and 10
Description: Blood pressure measurement included systolic blood pressure (SBP) and diastolic BP (DBP). Change in the mean blood pressure from Baseline was calculated as the post-Baseline value minus the Baseline value. Data are presented for change from Baseline at Day 1 (2 hours post dose [hrs]), Day 4 (1 hr pre-dose), Day 7 (1 hr pre-dose), and Day 10 (1 hr pre-dose and 2 hrs post dose).
Time Frame: Baseline and Days 1, 4, 7, and 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
millimeters of mercury (mmHg)
  SBP, Day 1, 2 hrs post dose | -5.93 (6.051) | -1.11 (6.348) | -2.17 (5.551) | 3.10 (12.927)
  SBP, Day 4, 1 hr pre-dose | -1.64 (10.221) | 1.78 (4.874) | 1.72 (11.880) | -7.60 (10.325)
  SBP, Day 7, 1 hr pre-dose | 0.08 (12.188) | -0.56 (10.227) | 2.28 (8.544) | -2.90 (9.351)
  SBP, Day 10, 1 hr pre-dose | -3.21 (11.419) | 2.89 (10.836) | 4.94 (6.640) | -6.40 (11.520)
  SBP, Day 10, 2 hrs post dose | -2.07 (11.193) | 2.67 (9.311) | 3.50 (10.974) | -6.40 (10.453)
  DBP, Day 1, 2 hrs post dose | 0.64 (5.321) | 1.39 (4.060) | 2.33 (4.183) | -2.70 (8.210)
  DBP, Day 4, 1 hr pre-dose | 0.50 (6.658) | 1.72 (7.480) | -0.67 (7.036) | -3.20 (4.423)
  DBP, Day 7, 1 hr pre-dose | -0.58 (7.262) | 1.61 (8.543) | 1.33 (6.708) | -2.40 (6.599)
  DBP, Day 10, 1 hr pre-dose | 0.07 (8.696) | 0.17 (4.690) | 4.11 (6.314) | -7.00 (7.619)
  DBP, Day 10, 2 hrs post dose | -0.79 (10.912) | 0.83 (8.775) | 6.00 (9.131) | -4.90 (8.140)

19. Primary Outcome: Change From Baseline in Mean Heart Rate at Days 1, 4, 7, and 10
Description: Heart rate is the measure of heart beats per minute (bpm). Change in the mean heart rate from Baseline was calculated as the post-Baseline value minus the Baseline value. Data are presented for change from Baseline at Day 1 (2 hours post dose [hrs]), Day 4 (1 hr pre-dose), Day 7 (1 hr pre-dose), and Day 10 (1 hr pre-dose and 2 hrs post dose).
Time Frame: Baseline and Days 1, 4, 7, and 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
beats per minute
  Day 1, 2 hrs post dose | -3.71 (6.861) | -7.67 (6.461) | -2.83 (5.734) | -6.85 (5.907)
  Day 4, 1 hr pre-dose | 3.43 (11.133) | -3.22 (6.610) | 6.50 (9.434) | 2.95 (12.513)
  Day 7, 1 hr pre-dose | 2.86 (10.984) | 0.67 (8.047) | 3.72 (8.511) | -2.85 (9.196)
  Day 10, 1 hr pre-dose | 3.29 (16.230) | 0.56 (9.547) | 3.83 (8.162) | -0.95 (8.268)
  Day 10, 2 hrs post dose | -1.57 (14.351) | 0.44 (13.907) | -3.72 (8.635) | -7.05 (7.890)

20. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: A 12-lead electrocardiogram (ECG) was performed by qualified personnel at the site after the participant had rested for at least 5 minutes in a semi-recumbent or supine position. If a QTc measurement of >=500 milliseconds (msec) was noted on a scheduled or unscheduled ECG, two additional ECGs were to be obtained within 5 minutes to confirm the abnormality. The number of participants with abnormal clinically significant (CS) and not clinically significant (NCS) ECG findings are presented here. The site determined if an ECG finding is significant or not. ECGs were obtained at Screening, Day 1 (pre-dose [twice] and then 1.0, 1.5, and 2.0 hours [hrs] post dose), Day 4 (pre-dose), Day 7 (pre-dose), Day 10 (pre-dose and then 1.0, 1.5, and 2.0 hrs post dose), Day 11 (prior to the 24 hr PK sample [pre lab]), and Follow-up.
Time Frame: Screening; Days 1, 7, 10, 11; and Follow-up (up to Study Day 21)
Population: Safety Population. Only those participants who were available at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
participants
  Screening, Normal, n=7, 9, 9, 10 | 5 | 7 | 8 | 9
  Screening, NCS, n=7, 9, 9, 10 | 2 | 2 | 1 | 1
  Screening, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 1, pre-dose 1, Normal, n=7, 9, 9, 10 | 5 | 7 | 9 | 8
  Day 1, pre-dose 1, NCS, n=7, 9, 9, 10 | 2 | 2 | 0 | 2
  Day 1, pre-dose 1, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 1, pre-dose 2, Normal, n=7, 9, 9, 10 | 5 | 7 | 9 | 8
  Day 1, pre-dose 2, NCS, n=7, 9, 9, 10 | 2 | 2 | 0 | 2
  Day 1, pre-dose 2, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 1, 1 hr post dose, Normal, n=7, 9, 9, 10 | 6 | 7 | 9 | 8
  Day 1, 1 hr post dose, NCS, n=7, 9, 9, 10 | 1 | 2 | 0 | 2
  Day 1, 1 hr post dose, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 1, 1.5 hrs post dose, Normal, n=7, 9, 9, 10 | 5 | 6 | 8 | 7
  Day 1, 1.5 hrs post dose, NCS, n=7, 9, 9, 10 | 2 | 3 | 1 | 3
  Day 1, 1.5 hrs post dose, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 1, 2 hrs post dose, Normal, n=7, 9, 9, 10 | 5 | 6 | 7 | 8
  Day 1, 2 hrs post dose, NCS, n=7, 9, 9, 10 | 2 | 3 | 2 | 2
  Day 1, 2 hrs post dose, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 4, pre-dose, Normal, n=7, 9, 9, 10 | 3 | 7 | 8 | 9
  Day 4, pre-dose, CS, n=7, 9, 9, 10 | 4 | 2 | 2 | 1
  Day 4, pre-dose, NCS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 7, pre-dose, Normal | 4 | 9 | 9 | 9
  Day 7, pre-dose, CS, n=7, 9, 9, 10 | 3 | 0 | 0 | 1
  Day 7, pre-dose, NCS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 10, pre-dose 1, Normal, n=7, 9, 9, 10 | 4 | 8 | 8 | 8
  Day 10, pre-dose 1, NCS, n=7, 9, 9, 10 | 3 | 1 | 1 | 2
  Day 10, pre-dose 1, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 10, 1 hr post dose, Normal, n=7, 9, 9, 10 | 4 | 7 | 8 | 8
  Day 10, 1 hr post dose, NCS, n=7, 9, 9, 10 | 3 | 2 | 1 | 2
  Day 10, 1 hr post dose, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 10, 1.5 hrs post dose, Normal, n=7, 9, 9, 9 | 2 | 7 | 8 | 8
  Day 10, 1.5 hrs post dose, NCS, n=7, 9, 9, 9 | 5 | 2 | 1 | 1
  Day 10, 1.5 hrs post dose, CS, n=7, 9, 9, 9 | 0 | 0 | 0 | 0
  Day 10, 2 hrs post dose, Normal, n=7, 9, 9, 10 | 3 | 7 | 8 | 7
  Day 10, 2 hrs post dose, NCS, n=7, 9, 9, 10 | 4 | 2 | 1 | 3
  Day 10, 2 hrs post dose, CS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Day 11, pre lab, Normal, n=7, 9, 9, 10 | 3 | 6 | 9 | 10
  Day 11, pre lab, CS, n=7, 9, 9, 10 | 4 | 3 | 0 | 0
  Day 11, pre lab, NCS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0
  Follow-up, Normal, n=7, 9, 9, 10 | 2 | 8 | 9 | 9
  Follow-up, CS, n=7, 9, 9, 10 | 5 | 1 | 0 | 1
  Follow-up, NCS, n=7, 9, 9, 10 | 0 | 0 | 0 | 0

21. Primary Outcome: Number of Participants With the Indicated Grade 3 and Grade 4 Laboratory Abnormalities
Description: Clinical laboratory toxicities were graded according to the National Institutes of Allergy and Infectious Diseases (NIAID), Division of Acquired Immunodeficiency Syndrome (DAIDS). Grade 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented only for Grade 3 and Grade 4 laboratory abnormalities. Clinical laboratory abnormalities included: increased glucose, lipase, decreased platelets, and triglycerides.
Time Frame: Screening; Days 1, 3, 7, and 10; and Follow-up (up to Study Day 21)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
participants
  Increased glucose, Screening, n=7, 9, 9, 10 | 0 | 1 | 0 | 0
  Increased Glucose, Day 7, n=7, 9, 9, 9 | 0 | 1 | 0 | 0
  Lipase, Day 10, n=7, 9, 9, 9 | 0 | 0 | 1 | 0
  Decreased platelets, Day 1, n=6, 9, 9, 9 | 0 | 0 | 1 | 0
  Decreased platelets, Day 3, n=6, 9, 9, 10 | 0 | 0 | 1 | 0
  Decreased platelets, follow-up, n=7, 9, 9, 10 | 0 | 0 | 1 | 0
  Triglycerides, Day 7, n=7, 9, 9, 9 | 0 | 0 | 1 | 0

22. Secondary Outcome: Median Change From Baseline in Plasma HIV-1 RNA Levels During the Follow-up Period (Days 11 to 21)
Description: Change from Baseline in Plasma HIV-1 RNA levels was calculated as the value during the Follow-up period minus the Basline value.
Time Frame: Baseline and Follow-up period (Days 11 to 21)
Population: ITT(E) Population
Measure: Median (Full Range); unit: Log10 copies/mL
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
Log10 copies/mL | -0.069 [-1.39 to 0.22] | -0.169 [-0.92 to 0.54] | -0.150 [-0.61 to 0.34] | -0.887 [-1.96 to 0.26]

23. Secondary Outcome: Mean Change From Baseline in Plasma HIV-1 RNA Levels During the Follow-up Period (Days 11 to 21)
Description: as for outcome 22
Time Frame: Baseline and Follow-up period (Days 11 to 21)
Population: ITT(E) Population
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
Log10 copies/mL | -0.188 (0.5443) | -0.149 (0.3931) | -0.154 (0.3126) | -0.899 (0.6997)

24. Secondary Outcome: Median Change From Baseline in Cluster of Differentiation 4+ (CD4+) Cell Count at Day 11
Description: Median change from Baseline in CD4+ cell count was calculated as the Day 11 value minus the Baseline value.
Time Frame: Baseline and Day 11
Population: Per-Protocol Population: all participants included in the ITT(E) Population, excluding those who had at least one major protocol deviation
Measure: Median (Full Range); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
Cells per cubic millimeter (cells/mm^3) | -28.5 [-247 to 50] | 15.0 [-286 to 222] | 106.0 [-39 to 142] | 64.0 [-155 to 523]

25. Secondary Outcome: Number of Participants With the Emergence of Drug Resistance Mutations
Description: The number of participants with the emergence (from Baseline) of drug resistance mutations at Day 11 was measured.
Time Frame: Baseline and Day 11
Population: ITT(E) Population
Measure: Number; unit: participants
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Number analyzed (Participants) | 7 | 9 | 9 | 10
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from Baseline (Day 1) until Follow-up (average of 3 study weeks).
Description: SAEs and non-serious AEs were collected in the Safety Population, comprised of all participants who were randomized into the study with documented evidence of having received at least one dose of randomized treatment.
Arm/Group | Placebo | GSK1349572 2 mg QD | GSK1349572 10 mg QD | GSK1349572 50 mg QD
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 5/7 | 4/9 | 7/9 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | GSK1349572 2 mg QD (N=9) | GSK1349572 10 mg QD (N=9) | GSK1349572 50 mg QD (N=10)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 2
Irritability (General disorders) | 1 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 2
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Daydreaming (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.